CLINICAL TRIAL: NCT03830203
Title: A Randomized, Double-Blind, Parallel-Group, Active-Control Study to Compare the Efficacy and Safety of BAT1806 to RoActemra® in Rheumatoid Arthritis Patients With Inadequate Response to Methotrexate
Brief Title: Comparative Study of BAT1806 to RoActemra® in Rheumatoid Arthritis Patients With Inadequate Response to Methotrexate
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-1806-002-CR
Record Dates: First submitted 2019-01-22; First posted 2019-02-05 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2020-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAT1806 (Experimental): BAT1806 injection: 8 mg/kg, intravenous infusion by 60 min
  Interventions: Drug: BAT1806
- Actemra(EU-licensed) (Active Comparator): Actemra(EU-licensed): 8 mg/kg, intravenous infusion by 60 min
  Interventions: Drug: Actemra(EU-licensed)

INTERVENTIONS:
Drug: BAT1806 — 8 mg/kg
  Arms: BAT1806
Drug: Actemra(EU-licensed) — 8 mg/kg
  Arms: Actemra(EU-licensed)

SUMMARY:
This is a Phase 3, multicenter, multinational, randomized, double-blind, parallel-group, active-control study to compare efficacy, safety, immunogenicity, and PK of BAT1806 compared with RoActemra in subjects with RA that is inadequately controlled by MTX.

The study is composed of a ≤ 28-day screening period, a 24-week initial treatment period (TP1), a 24 week secondary treatment period (TP2), and an extra 4-week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age or older who fulfil the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) 2010 revised classification criteria for RA diagnosis for at least 6 months before screening, based on the medical history record.
2. Subject presents with active RA, as defined by:

   1. ≥ 6 out of 68 tender joints (at screening and randomization) AND
   2. ≥ 6 out of 66 swollen joints (at screening and randomization) AND
   3. Serum C-reactive protein (CRP) > upper limit of normal (ULN) value or erythrocyte sedimentation rate (ESR) ≥ 28 mm/hour at screening.
3. Subjects are eligible if they have received not more than 2 biological agents other than interleukin-6 inhibitors or targeted synthetic DMARDs (eg, tofacitinib) in total for RA treatment.
4. Female subjects of childbearing potential and male subjects with a female partner of childbearing potential must be willing to take reliable contraceptive precautions throughout the study period and continuing for at least 3 months after the last dose of study drug. Reliable methods of contraception include: intrauterine device, hormonal contraceptives (eg, oral, patch, or injectable), male vasectomy (if vasectomy was medically confirmed), a barrier protection method (eg, condom or diaphragm) in association with spermicide cream, foam, or gel. Abstinence from heterosexual intercourses is accepted when this is the usual lifestyle of the subject and must be continued for at least 3 months after the last dose of study drug. A female subject is considered not of child-bearing potential when postmenopausal (at least 12 consecutive months without menses without an alternative medical cause) or surgically sterilized (bilateral tubal ligation, bilateral oophorectomy with or without hysterectomy).
5. If female of childbearing potential, subject should have a negative pregnancy test result at screening and baseline visit.
6. Subjects must be willing to provide written consent and to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Has RA of ACR functional class IV or is wheelchair/bed bound.
2. Known hypersensitivity to tocilizumab or to study treatment excipients.
3. Subject has received any cell-depleting therapy (eg, rituximab) ≤ 12 months prior to randomization.
4. Subject has been treated with an investigational drug other than those prohibited or device ≤ 8 weeks or 5 half-lives of the drug (whichever is longer) prior to randomization.
5. Subject has undergone joint surgery ≤ 12 weeks prior to randomization (on any joint to be assessed during the study) or has any surgery planned during the study.
6. Evidence of malignancy, lung infection, or abnormalities suggestive of active tuberculosis (TB) on chest radiography performed within 12 weeks prior to the Screening Visit or during the screening period.
7. Any recurrent bacterial, fungal, or viral infection that based on the investigator´s clinical assessment makes the subject unsuitable for the study, including recurrent/disseminated herpes zoster.
8. Current or history of diverticulitis, complications of diverticulitis, history of diverticulosis requiring antibiotic treatment, current or history of chronic ulcerative lower gastrointestinal tract diseases or any other lower gastrointestinal condition that may predispose to perforation.
9. Any history of malignancy or lymphoproliferative disease at any time, except curative treatment for nonmelanoma skin cancer or resected carcinoma in situ of the cervix.
10. Have a transplanted organ/tissue or stem cell transplantation.
11. Subject has an underlying metabolic, hematologic, renal, hepatic, pulmonary, neurologic, endocrine, cardiac, infectious, or gastrointestinal condition, which in the opinion of the investigator places the subject at unacceptable risk.
12. Subject has a history of demyelinating diseases (including myelitis) or neurologic symptoms suggestive of demyelinating disease.
13. Subject has received any live or attenuated vaccine ≤ 4 weeks prior to randomization or plans to receive it during the study including the safety follow up period.
14. Subject has a history of clinically significant drug or alcohol abuse in the last 12 months as judged by the investigator.
15. Pregnant or nursing (lactating) women.
16. Subject is considered by the investigator, for any reason, to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 621 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-01-05 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With an American College of Rheumatology 20 Percent (%) (ACR20) Response | 6 months
  ACR20 response, ≥ 20 percent (%) improvement in tender joint count; ≥ 20% improvement in swollen joint count; and = at least 20% improvement in at least 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant (ESR).

SECONDARY OUTCOMES:
Change From Baseline in DAS28 | 1 year
  The DAS28 is a score on a scale (0 to 10) indicating current activity of rheumatoid arthritis (>5.1=high disease activity; <=3.2=low disease activity; <2.6=remission); a continuous variable which is a composite of 4 variables (the number of tender joints out of 28, the number of swollen joints out of 28 joints, erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]) and patient's global assessment (PGA) of disease activity measured on a visual analogue scale (VAS) of 100 mm). Change equals (=) Week X observation minus (-) Baseline observation.

OTHER OUTCOMES:
Percentage of Participants With an ACR20 Response | 1 year
  ACR20 response, ≥ 20 percent (%) improvement in tender joint count; ≥ 20% improvement in swollen joint count; and = at least 20% improvement in at least 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and acute phase reactant (ESR).
Percentage of Participants With an ACR50 Response | 1 year
  ACR50 response: ≥ 50% improvement in tender joint count; = ≥50% improvement in swollen joint count; and = at least 50% improvement in 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and acute phase reactant (ESR).
Percentage of Participants With an ACR70 Response | 1 year
  ACR70 response: ≥ 70% improvement in tender joint count; = ≥70% improvement in swollen joint count; and = at least 70% improvement in 3 of the following 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and acute phase reactant (ESR).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zeng, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ebbers HC, Taylor PC, Leng X, Wei W, Kinsella NM, Zhou Y, Yang X, Chamberlain P. A Comparison of the Immunogenicity of Intravenous BAT1806, a Tocilizumab Biosimilar, and Its Reference Product. Rheumatol Ther. 2025 Jun;12(3):529-546. doi: 10.1007/s40744-025-00760-y. Epub 2025 Apr 8. PMID 40198544
- [Derived] Leng X, Leszczynski P, Jeka S, Liu S, Liu H, Miakisz M, Gu J, Kilasonia L, Stanislavchuk M, Yang X, Zhou Y, Dong Q, Mitroiu M, Addison J, Rezk MF, Zeng X. A phase 3, randomized, double-blind, active-controlled clinical trial to compare BAT1806/BIIB800, a tocilizumab biosimilar, with tocilizumab reference product in participants with moderate-to-severe rheumatoid arthritis with inadequate response to methotrexate: treatment period 2 analysis (week 24 to week 48). Arthritis Res Ther. 2024 Sep 7;26(1):157. doi: 10.1186/s13075-024-03375-w. PMID 39244595
- [Derived] Leng X, Leszczynski P, Jeka S, Liu SY, Liu H, Miakisz M, Gu J, Kilasonia L, Stanislavchuk M, Yang X, Zhou Y, Dong Q, Rezk M, Mitroiu M, Addison J, Zeng X. Comparing tocilizumab biosimilar BAT1806/BIIB800 with reference tocilizumab in patients with moderate-to-severe rheumatoid arthritis with an inadequate response to methotrexate: a phase 3, randomised, multicentre, double-blind, active-controlled clinical trial. Lancet Rheumatol. 2024 Jan;6(1):e40-e50. doi: 10.1016/S2665-9913(23)00237-0. PMID 38258678